CLINICAL TRIAL: NCT05475301
Title: Incidence, Risk Factor, Treatment and Overall Survival of Locally Recurrent Rectal Cancer: a Retrospective, Population-based Cohort Study
Brief Title: Incidence, Risk Factor, Treatment and Overall Survival of Locally Recurrent Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Hidde Swartjes, Researcher in training, Radboud University Medical Center
Other Study IDs: K20.256
Record Dates: First submitted 2022-07-15; First posted 2022-07-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Rectal Neoplasms; Neoplasm Recurrence, Local
MeSH Terms: conditions — Rectal Neoplasms; Neoplasm Recurrence, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data on disease recurrence was collected for all primary rectal cancer patients diagnosed in the Netherlands over the first six months of 2015. Three-year cumulative incidence, risk factors, treatment and three-year OS of locally recurrent rectal cancer were determined.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage I-III primary rectal carcinoma;
* Diagnosed between January 1st and June 30th of 2015;
* TME resection of primary rectal carcinoma.

Exclusion Criteria:

* Neuroendocrine tumor morphology;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with stage I-III primary rectal cancer in the first half of 2015.
Sampling Method: Non-Probability Sample
Enrollment: 1431 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of patients with locally recurrent rectal cancer in curatively treated primary rectal cancer patients | Three years
  UNIT OF MEASUREMENT: Cumulative incidence of patients with locally recurrent rectal cancer in curatively treated primary rectal cancer patients MEASUREMENT TOOL: Registration of diagnosis of locally recurrent rectal cancer in the electronic patient file.
  The competing-risk cumulative incidence will be calculated, which will inform on the proportion of patients who have developed locally recurrent rectal cancer at that time point.
Risk factors for development of locally recurrent rectal cancer in curatively treated primary rectal cancer patients | Three years
  UNIT OF MEASUREMENT: Risk factors for development of locally recurrent rectal cancer in primary rectal cancer patients MEASUREMENT TOOL: Registration of clinical and pathological covariates of primary rectal cancer in the electronic patient file and national pathological database (PALGA).
  Clinical and pathological risk factors for the development of locally recurrent rectal cancer will be identified using multivariable competing-risk risk regression analyses, according to the cause-specific hazard approach. This will inform on specific clinical and pathological covariates which increase or decrease the risk for development of locally recurrent rectal cancer.
Proportions of treatment given to patients with locally recurrent rectal cancer | Three years
  UNIT OF MEASUREMENT: Proportions of treatment given to patients with locally recurrent rectal cancer; MEASUREMENT TOOL: Registration of treatment for locally recurrent rectal cancer in the electronic patient file.
  Using descriptive statistics, treatment patterns of patients with locally recurrent rectal cancer will be identified. Groups that will be created, will also be used to assess overall survival.
Overall survival of patients with locally recurrent rectal cancer | Three years
  UNIT OF MEASUREMENT: Overall survival of patients with locally recurrent rectal cancer; MEASUREMENT TOOL: Registration of vital status in the national personal records database.
  Overall survival will be estimated for patients with locally recurrent rectal cancer, stratifying for different groups (i.e. treatment, diagnosis of synchronous metastases, diagnosis within first year after primary resection, etc.)

IPD SHARING:
Plan to Share IPD: No
Data can be requested through the Netherlands Cancer Registry.